CLINICAL TRIAL: NCT03112265
Title: Using Neuroimaging to Understand Children's Mental Health and Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Professor and Primary Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 313704
Record Dates: First submitted 2017-03-28; First posted 2017-04-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Depression; Trauma; Behavior Problems
Keywords: anxiety; depression; trauma; behavior problems; evidence-based treatments; manualized treatments; cognitive-behavioral therapy; youth; mental health; self-regulation; neuroimaging
MeSH Terms: conditions — Anxiety Disorders; Depression; Wounds and Injuries; Mental Disorders; Psychological Well-Being; Self-Control | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Child STEPS (Experimental): Child STEPs includes (1) a treatment protocol, Modular Approach to Therapy for Children with Anxiety, Depression, Trauma or Conduct Problems (MATCH-ADTC), and (2) a youth monitoring and feedback system (MFS).
  Interventions: Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems; Other: Monitoring and Feedback System
- Usual Care (Active Comparator): Treatment in the UC condition will use the procedures therapists and their supervisors consider appropriate and believe to be effective, and researchers will not influence their work.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems — MATCH-ADTC is designed for children aged 6-15. Unlike most evidence-based treatments (EBTs), which focus on single disorder categories (e.g., anxiety only), MATCH is designed for multiple disorders and problems encompassing anxiety, depression, post-traumatic stress, and disruptive conduct, including the conduct problems associated with ADHD. MATCH is composed of 33 modules-i.e., specific treatment procedures derived from decades of research on EBTs. The various modules can be organized and sequenced flexibly to tailor treatment to each child's characteristics and needs.
  Other Names: MATCH; MATCH - ADTC
  Arms: Child STEPS
Other: Monitoring and Feedback System — For each child, the web-based MFS system provides weekly monitoring of the MATCH modules used and the child's treatment response, in two forms (a) changes on the Behavior and Emotions Survey and (b) changes in severity of the top treatment concerns identified by youths and caregivers. At the end of treatment, the MFS provides a complete record of modules used, and child treatment response, across all the weeks of treatment.
  Other Names: MFS
  Arms: Child STEPS
Behavioral: Treatment as usual — Treatment in the UC condition will use the procedures therapists and their supervisors consider appropriate and believe to be effective.
  Other Names: Usual Care; UC
  Arms: Usual Care

SUMMARY:
The study will compare the impact of Child STEPs versus usual school-based therapy on neural and companion behavioral measures of self-regulation.

DETAILED DESCRIPTION:
This project will implement and evaluate the Child STEPs treatment approach as compared to "treatment as usual" (known as Usual Care or UC) through a randomized controlled trial (RCT) at eight K-8 public schools. The STEPs model has two components: (1) a modular protocol that combines 33 modules-i.e., descriptions of common elements within evidence-based therapies for anxiety, depression, post-traumatic stress, and conduct problems; and (2) a web-based system for monitoring student responses to treatment and providing weekly feedback to therapists to guide their selection and sequencing of the STEPs modules. The project will examine: (a) whether self-regulation skills at baseline are associated with baseline patterns of mental health and school problems; (b) whether self-regulation skills at baseline predict degree of improvement during treatment; (c) whether self-regulation skills improve from pre-to post treatment, and whether extent of this improvement differs by treatment condition; and (d) whether self-regulation improvement (from pre-to-post treatment) mediates the long-term benefit of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. enrolled in grades 3-7
2. have a primary clinical problem in the areas of anxiety, depression, conduct, or posttraumatic stress
3. clinically elevated problem levels on the Internalizing, Externalizing, Anxious-Depressed, Withdrawn-Depressed, Aggressive Behavior, or Rule-Breaking Behavior scales of the Child Behavior Checklist or Youth Self-Report or on the UCLA Post-Traumatic Stress Disorder Reaction Index.

Exclusion Criteria:

1. Mental retardation
2. Pervasive developmental disorder
3. Eating disorder
4. children for whom attention problems or hyperactivity are the primary referral concern
5. active psychosis and/or a suicide attempt in the previous year

To participate in the two neuroimaging tasks (Emotion Regulation Task; Emotional Go/No Go Task), participants must be healthy (no major medical illness), right-handed, fluent in English, have no history of neurological impairment (including but not limited to history of loss of consciousness for great than 20 minutes, seizures, stroke, etc.), have normal or corrected to normal vision, and have no contra-indications or risk factors for MRI research (such as braces or metal implants).

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Emotion Regulation Task at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Emotional Go/No-Go Task at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks

SECONDARY OUTCOMES:
Change from Baseline Attentional Bias Task at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Granularity Task at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Behavior Rating Inventory of Executive Function (BRIEF) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Early Adolescent Temperament Questionnaire Revised (EATQ-R) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks

OTHER OUTCOMES:
Change from Baseline Coping with Children's Negative Emotions Scale (CCNES) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Parenting Stress Index-Short Form (PSI-SF) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Family Adaptability and Cohesion Scale IV (FACES-IV) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks
Change from Baseline Five Minute Speech Sample (FMSS) at End of Treatment | Change over time from Day 1 to end of treatment, assessed up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John R. Weisz, PhD, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Weisz JR, Chorpita BF, Palinkas LA, Schoenwald SK, Miranda J, Bearman SK, Daleiden EL, Ugueto AM, Ho A, Martin J, Gray J, Alleyne A, Langer DA, Southam-Gerow MA, Gibbons RD; Research Network on Youth Mental Health. Testing standard and modular designs for psychotherapy treating depression, anxiety, and conduct problems in youth: a randomized effectiveness trial. Arch Gen Psychiatry. 2012 Mar;69(3):274-82. doi: 10.1001/archgenpsychiatry.2011.147. Epub 2011 Nov 7. PMID 22065252
- [Background] Chorpita, B.F., & Weisz, J.R. (2009). Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH-ADTC). Satellite Beach, FL: PracticeWise, LLC.